CLINICAL TRIAL: NCT03014349
Title: Water Drinking Test and Its Reproducibility in Goldmann Applanation Tonometry and Pneumatic Tonometry
Acronym: WDTRGP
Status: Completed | Type: Observational
Sponsor: VER Excelência em Oftalmologia (Other)
Responsible Party: Principal Investigator, Rodrigo Egidio da Silva, ophthalmologist, VER Excelência em Oftalmologia
Other Study IDs: VEREO
Record Dates: First submitted 2016-12-09; First posted 2017-01-09 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Glaucoma Suspect
Keywords: Glaucoma; Ocular hypertension
MeSH Terms: conditions — Ocular Hypertension; Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- primary open-angle glaucoma and/or glaucoma suspects: Individuals with primary open-angle glaucoma and/or glaucoma suspects, selected from the electronic records of the VER Hospital. The following variables will be observed: gender, age, race, systemic diseases, intraocular pressure, type of glaucoma, complementary exams and degree of evolution. All patients were given a complete ophthalmologic examination, including Goldmann and pneumatic tonometry.
  Interventions: Other: Analysis of medical records

INTERVENTIONS:
Other: Analysis of medical records — Individuals with primary open-angle glaucoma and/or glaucoma suspects, selected from the electronic records of the VER Hospital. The following variables will be observed: gender, age, race, systemic diseases, intraocular pressure, type of glaucoma, complementary exams and degree of evolution. All patients were given a complete ophthalmologic examination, including Goldmann and pneumatic tonometry.

SUMMARY:
The purpose of this study is to evaluate the reproducibility of tonometry in the Goldmann applanation apparatus and pneumatic in the water drinking test.

DETAILED DESCRIPTION:
Glaucoma consists of a multifactorial disease caused by a deficiency in drainage of the aqueous humor, which may cause an increase in intraocular pressure (IOP), an impairment of the optic nerve and visual field changes. According to the most recent data , this disease is the second cause of blindness in the world (12.3%). An estimate indicates that, by 2020, there will be 79.6 million glaucomatous individuals in the world. The estimated prevalence of primary glaucoma in the Brazilian population was 3.4%, consisting of 2.4% open angle and 0.7% closed angle.

Glaucoma can be: open angle, angle-closure, congenital or secondary. Increased IOP is the major risk factor for glaucoma progression as well as its fluctuation (difference between the highest and lowest IOP measure) in primary open-angle glaucoma (POAG). In addition, age, family history, central corneal thickness, race, high myopia, hypermetropia, diabetes mellitus, hypertension and hypotension, gender, optic disc hemorrhages, suspected optic nerve excavation, and cardiovascular and cerebrovascular diseases.

The treatment depends on the classification of glaucoma, since in the POAG, the initial treatment is with topical monotherapy (ocular hypotensors). However, in some situations, drug treatment is not enough to stabilize the process of glaucomatous progression. In these cases, incisional surgery or laser treatment is necessary.

Trabeculectomy consists of an intervention to increase drainage of the aqueous humor, in order to control the IOP and prevent the progression of the disease. However, due to its complications, such as atalamia, hypotonia, the development of cataract and the risk of endophthalmitis, this procedure is indicated in the refractory cases to clinical and/or laser treatment. Thus, clinical treatment and trabeculoplasty are the treatments of choice. Trabeculoplasty is indicated in the cases of POAG, pseudoexfoliative, pigmented and in some cases of secondary and trabecular glaucoma visible to the gonioscopy.

The tonometer is the device used to detect IOP increase. Despite the existence of several models, Goldmann's applanation is considered the gold standard for this measurement, since it evaluates the force necessary to deform the surface of the cornea. This method is quite accurate, however, errors may occur in the result due to fluorescein patterns, very thick corneas, excessive pressure on the eyeball when holding the patient's eyelids or elevated corneal astigmatism without the adequate compensatory positioning of the planer.

The measurement of IOP can also be performed through another type of tonometer: non-contact, pneumatic or blow. It was first used in 1973 by Forbes and its advantages are: 1) no need for the use of eye drops, 2) it can be performed by people who are not doctors, 3) it has a low risk of contamination and 4) it can be used for screening programs. However, a study by Britt et al. showed the presence of lachrymal film dehiscence and the existence of microaerosol with the air blow, which would make this method not so aseptic.

According to the study, where the pneumatic tonometer was compared with that of Goldmann, the results obtained were: 50% of the evaluated eyes showed no differences between the two devices and in 85% they were between approximately 2 mmHg. In another study which compared the IOP values measured by the mentioned tonometers, it was verified that the pneumatic tonometer underestimates the IOP values, compared to Goldmann, in thin corneas; however, there is no significant difference between the measurements of the two tonometers in thick corneas.

The Water Drinking Test (WDT) is a propaedeutic widely used to evaluate the maximum intraocular pressure (IOP) and its fluctuation. These data are extremely important for the expected result in relation to the reproducibility of the exams, since in the study , showed that the WDT can be used to estimate the peak and diurnal fluctuation of supine IOP in the simplified daily stress curve (another method for the same purpose of the WDT) in patients under treatment for glaucoma.

Glaucoma is a serious eye health problem, as it has a high incidence and prevalence worldwide and is the leading cause of irreversible blindness in the world. Therefore, it is extremely important to perform tests that will detect altered IOP values.

The IOP values obtained over a 24 hour period are important data, since they are required to control and conduct the treatment of glaucoma. In the past, the WDT has often been used to diagnose patients with this pathology. Due to a series of studies,it was found that the WDT can not be used as a diagnostic test, but as a tool to evaluate changes in IOP peaks. In addition, a comparison of reproducibility between devices will facilitate a better evaluation, speed, safety and efficacy in the treatment, contributing to increase the quality of life of the patient and also to guide other studies in this area.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Intraocular pressure greater than 21 mmhg
* Optic neuropathy more than 0.5
* CampimetryPerimetric suggestive of glaucoma

Exclusion Criteria:

* Were patients under 18 years of age
* Incomplete data in electronic records
* Had previous ophthalmologic surgeries or other non-glaucoma-related ophthalmic diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of individuals with primary open-angle glaucoma and/or glaucoma suspects
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Water drinking test and its reproducibility in Goldmann applanation tonometry | Six months
Water drinking test and its reproducibility in pneumatic tonometry | Six months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wachtl J, Toteberg-Harms M, Frimmel S, Kniestedt C. [Evaluation of correction formulas for tonometry : The Goldmann applanation tonometry in approximation to dynamic contour tonometry]. Ophthalmologe. 2017 Aug;114(8):716-721. doi: 10.1007/s00347-016-0409-3. German. PMID 27921133
- [Background] Sakata R, Aihara M, Murata H, Saito H, Iwase A, Yasuda N, Araie M. Intraocular pressure change over a habitual 24-hour period after changing posture or drinking water and related factors in normal tension glaucoma. Invest Ophthalmol Vis Sci. 2013 Aug 7;54(8):5313-20. doi: 10.1167/iovs.13-11792. PMID 23821194
- [Background] Medina FM, Rodrigues FK, Filho Pde T, Matsuo T, Vasconcellos JP, Costa VP. Reproducibility of water drinking test performed at different times of the day. Arq Bras Oftalmol. 2009 May-Jun;72(3):283-90. doi: 10.1590/s0004-27492009000300002. PMID 19668954
- [Background] Meirelles SH, Yamane R, Alvares RM, Botelho PB, Morais FB, Moreira PB, Dantas AM, de Moraes Junior HV. [Comparative study between diurnal intraocular pressure curve and the association of ambulatory intraocular pressure curve with the water-drinking test in open angle glaucoma, normal tension glaucoma and normal eyes]. Arq Bras Oftalmol. 2007 May-Jun;70(3):471-9. doi: 10.1590/s0004-27492007000300015. Portuguese. PMID 17768555
- [Background] Medeiros FA, Sample PA, Zangwill LM, Bowd C, Aihara M, Weinreb RN. Corneal thickness as a risk factor for visual field loss in patients with preperimetric glaucomatous optic neuropathy. Am J Ophthalmol. 2003 Nov;136(5):805-13. doi: 10.1016/s0002-9394(03)00484-7. PMID 14597030
- [Background] Caiado RR, Badaro E, Kasahara N. Intraocular pressure fluctuation in healthy and glaucomatous eyes: a comparative analysis between diurnal curves in supine and sitting positions and the water drinking test. Arq Bras Oftalmol. 2014 Oct;77(5):288-292. doi: 10.5935/0004-2749.20140073. Epub 2014 Sep 1. PMID 25494373
- [Background] Regev G, Harris A, Siesky B, Shoshani Y, Egan P, Moss A, Zalish M, WuDunn D, Ehrlich R. Goldmann applanation tonometry and dynamic contour tonometry are not correlated with central corneal thickness in primary open angle glaucoma. J Glaucoma. 2011 Jun-Jul;20(5):282-6. doi: 10.1097/IJG.0b013e3181e66498. PMID 20577097
- [Background] Guler M, Bilak S, Bilgin B, Simsek A, Capkin M, Hakim Reyhan A. Comparison of Intraocular Pressure Measurements Obtained by Icare PRO Rebound Tonometer, Tomey FT-1000 Noncontact Tonometer, and Goldmann Applanation Tonometer in Healthy Subjects. J Glaucoma. 2015 Oct-Nov;24(8):613-8. doi: 10.1097/IJG.0000000000000132. PMID 25264986
- [Background] Quaranta L, Konstas AG, Rossetti L, Garcia-Feijoo J, O'Brien C, Nasr MB, Fogagnolo P, Demos CM, Stewart JA, Stewart WC. Untreated 24-h intraocular pressures measured with Goldmann applanation tonometry vs nighttime supine pressures with Perkins applanation tonometry. Eye (Lond). 2010 Jul;24(7):1252-8. doi: 10.1038/eye.2009.300. Epub 2009 Dec 4. PMID 19960033